CLINICAL TRIAL: NCT00867243
Title: Prediction of Hepatitis C Recurrence in Liver Transplant Recipients
Status: Terminated | Type: Observational
Why Stopped: This project is no longer being adequately supported to allow completion
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, TBaker, Assitant Professor of Surgery, Division of Organ Transplantation, Dept of Surgery, Northwestern University
Other Study IDs: STU12442 1963-002
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Complication of Transplanted Liver; Hepatitis C, Chronic
Keywords: Hepatitis C virus; HCV; Hepatitis C (and cirrhosis); Liver cirrhosis not due to HCV infection
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Recipient specimens: Peripheral blood draws at baseline and follow-up clinic visits.
  Donor specimens: Donor cells will be isolated from lymph nodes obtained at time of harvest; if living donor - blood taken at time of liver resection surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: HCV Positive: 50 patients whom are HCV positive
- Group 2: HCV Negative: 50 patients whom are HCV negative.

SUMMARY:
The purpose of the study is to look at cells of the immune system to see if the cells are different among people with different risk factors that have received a liver transplant. We will enroll 50 patients receiving liver transplant and their donors. Both donor and recipient must participate in the order for the recipient to participate in the study. We will take blood samples from these patients and their donors.

DETAILED DESCRIPTION:
To establish whether in-vitro donor-specific immune reactivity patterns can differentiate between those liver transplant recipients who are positive for the Hepatitis C virus (HCV) who are at high risk and those who are at low risk for graft loss secondary to early recurrence of HCV.

An assessment of the recipient's donor-specific immune status can be achieved by measuring T-cell activity, specifically alloreactive primed (donor-specific) T cell activity. It has been shown that detection of IFN-y in short-term enzyme-linked-immunosorbent-spot (ELISPOT) assay is consistent with the presence of primed memory T cells (6). In the transplantation setting, T cells of an allograft recipient that secret IFN-y after short in-vitro exposure to donor cells represent a prior sensitization of recipient to donor antigens in vivo. Clinically interpreted - this priming event may signify the presence of an up-coming, or an on-going, rejection episode. Our limited preliminary data suggest an additional potential clinical value for the in-vitro assessment of donor-specific IFN-y production in predicting those liver transplant recipients at higher risk for recurrence of Hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >18 years of age
* Chronic HCV infection (and cirrhosis) - group 1
* HCV RNA positive pre-transplant - group 1
* Liver cirrhosis not due to HCV infection - group 2

Exclusion Criteria:

* All patients < than 18 years of age
* Patients with hepatitis C infection
* Candidates receiving multi-organ combined transplantation
* Patients who have received a previous liver transplantation
* Patients who are unable to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is males/females over the age of 18 that require liver transplantation, and their donors
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2005-10; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To assess whether in-vitro donor-specific immune reactivity patterns are indicative of rate of HCV recurrence | Baseline prior to surgery, Weeks 1, 2; Months 1, 2, 3, 4, 5, 6, 12, 18

SECONDARY OUTCOMES:
To compare in-vitro donor-specific immune reactivity patterns and rejection episodes in liver transplant recipients | Baseline prior to surgery, Weeks 1, 2; Months 1, 2, 3, 4, 5, 6, 12, 18
To establish immune monitoring protocol for HCV+ liver transplant recipients that will aid in tailoring immunosuppression protocols for these patients and in devising strategies to treat patients with recurrent hepatitis C post-liver transplantation. | Baseline prior to surgery, Weeks 1, 2; Months 1, 2, 3, 4, 5, 6, 12, 18

CONTACTS AND LOCATIONS:
Overall Officials: Talia Baker, MD, Principal Investigator — Northwestern Memorial Hospital; Anat Tambur, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Tambur AR, Ben-Ari Z, Herrera ND, Klein T, Michowiz R, Mor E. Donor-specific hyporesponsiveness in ELISPOT assay is associated with early recurrence of hepatitis C in liver transplant recipients. Hum Immunol. 2005 Jan;66(1):21-7. doi: 10.1016/j.humimm.2004.08.180. PMID 15620458